CLINICAL TRIAL: NCT03886350
Title: Implication of UNconventionaL T Lymphocytes in Cystic Fibrosis
Brief Title: Implication of UNconventionaL T Lymphocytes in Cystic Fibrosis (UNLOCk)
Acronym: UNLOCk
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI18 / UNLOCk; 2019-A00290-57 (Other: IdRCB)
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Cystic Fibrosis; Innate Immunity; Inflammatory Response
Keywords: Unconventional T cells; Cystic fibrosis; gamma delta T cell; Mucosal Associated Invariant T cell; Natural Killer T cell
MeSH Terms: conditions — Cystic Fibrosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples Sputum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with cystic fibrosis: Patients with CF whom follow-up is undertaken at University Hospital of Tours, France
  Interventions: Other: blood and sputum samples

INTERVENTIONS:
Other: blood and sputum samples — Blood and sputum samples for research purpose collected during routine tests performed at steady state and acute exacerbation

SUMMARY:
Cystic fibrosis (CF) is characterized by a decrease in mucociliary clearance, recurrent infections and airway inflammation. This inflammatory process in airway mucosa is persistent, uncontrolled, but, somewhat paradoxically, ineffective for pathogen clearance. Neutrophils are chronically recruited in the airway mucosa by proinflammatory mediators such as Interleukin (IL)-17. However, mechanisms involved in this dysregulated and persistent immune response are not well understood.

In this context, a heterogeneous subpopulation of T lymphocytes called "unconventional T cells" (UTC) should deserve greater attention. UTC play a key role in orchestrating the ensuing innate and adaptive immune responses and they are endowed with numerous regulatory and effector properties. UTC mainly establish residency at mucosal sites, including the lung. To date, however, data related to implication and behavior of UTC during cystic fibrosis are extremely limited.

The hypothesis is that, given UTC properties, their functions and behavior are altered in CF, and thus, these cells could be implicated in persistent inflammation and poor response to infections.

The objective is to study UTC properties and functions in cystic fibrosis using blood and sputum samples of patients with CF, in correlation with comprehensive clinical and microbiological data.

The study will enroll adult patients with CF followed-up at University Hospital of Tours, France. For each patient included, blood and sputum samples will be analyzed during 18 months 1/ from routine tests obtained at steady state and 2/ from tests performed during acute exacerbations. UTC will be explored in blood and sputum using flowcytometry approach, to evaluate their relative abundance, activation/inhibition profile and functions (cytokine production and cytotoxic ability). Correlation will be made with clinical status, with longitudinal comparison across the study period for each patient, and comparison with the other patients and healthy volunteers.

This study will add significant knowledge in CF immunopathology by comprehensively assess UTC presence, functions and activation in CF. Indeed, UTC could be explored for disease progression marker, and, in a long-term perspective, explored for therapeutic interventions aiming at modulating their function (by activating or inhibiting UTC), to reshape lung immune response during CF.

DETAILED DESCRIPTION:
- Clinical and scientific background

Cystic fibrosis is characterized by functional abnormalities in the cystic fibrosis transmembrane conductance regulator (CFTR) membrane channel leading to a decrease in mucociliary clearance, recurrent infections and airway inflammation. This inflammatory process in airway mucosa is persistent, uncontrolled, but, somewhat paradoxically, ineffective for pathogen clearance. Neutrophils are chronically recruited in the airway mucosa by proinflammatory mediators such as IL-17, and probably largely contribute to tissue damage. However, up-stream mechanisms involved in this dysregulated and persistent immune response are not well understood.

In this context, seeking for new candidates that may be involved in this chronic inflammation is critical as there is, to date, no effective treatment to modulate immune response in CF. To address this, a heterogeneous subpopulation of T lymphocytes called "unconventional T cells" (UTC) should deserve greater attention. These cells comprise Natural Killer T (NKT) cells, mucosal associated invariant T cells (MAIT cells) and γδ T cells. The investigators believe these cells could be instrumental for future immune-intervention in CF immunopathology. First, UTC play a key role in orchestrating the ensuing innate and adaptive immune responses. Their pivotal role in mounting host defense during infection have been demonstrated, by the investigators and others, in different experimental models. Notably, their pivotal role for IL-17-driven neutrophil recruitment during acute pulmonary infection is well documented. Second, they are endowed with numerous regulatory and effector properties. Third, UTC mainly establish residency at mucosal sites, including the lung. Last, these cells are already investigated for therapeutic interventions (mainly in oncology, with ongoing phase I and II clinical trials). To date, however, data related to implication and behavior of UTC during cystic fibrosis are extremely limited and preliminary.

The hypothesis is that, given UTC properties, their functions and behavior are altered in CF, and thus, these cells could be implicated in persistent inflammation and poor response to infections.

- Objective of the study: The objective is to study UTC properties and functions in cystic fibrosis using blood and sputum samples of patients with CF, in correlation with comprehensive clinical and microbiological data.

- Design:

This is a prospective exploratory single-center study including adult patients with CF whom follow-up is undertaken at University Hospital of Tours, France.

Number of participants: 80

- Interventions and analysis:

For each patient included, study duration will be 18 months, during which blood and sputum samples will be analyzed 1/ from routine tests obtained at steady state during annual check-up and follow-up examination and 2/ from tests performed during acute exacerbations treated at the hospital or outpatient. To be enrolled in this study does not add any medical or biological examination compared to the usual follow-up. Each blood or sputum test done during follow-up examination or treating care will lead to supplementary samples for research.

Clinical parameters will be collected including clinical status (exacerbation or not), microbial status, pulmonary function test, drugs used like CFTR modulator therapies (lumacaftor ivacaftor) or antibiotics.

UTC will be explored in blood and sputum using flowcytometry approach, to evaluate their relative abundance, activation/inhibition profile and functions (cytokine production and cytotoxic ability). In some cases, intra-cellular staining will be performed to assess cytokine production and/or transcription factor expression. Functions of unconventional T cells will also be performed after ex vivo stimulation on purified population (cell sorting). Cytokine level sand transcriptomic analyses will also be performed on blood samples.Correlation will be made with clinical status, with longitudinal comparison across the study period for each patient, and comparison with the other patients and healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a genetic diagnosis of cystic fibrosis
* Older than 18 years old
* Be followed-up at University Hospital of Tours

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patient under judicial protection
* Patient having objected to the processing of his data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with cystic fibrosis whom follow-up is undertaken at University Hospital of Tours.
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Blood level of Non-Conventional T Lymphocytes | 18 months
  Blood UTC expressed as % Cluster of Differenciation 3+ (CD3+) lymphocytes (gamme delta T lymphocytes, MAIT cells, Natural Killer T cells)
Sputum level of Non-Conventional T Lymphocytes | 18 months
  Sputum UTC expressed as % CD3+ lymphocytes (gamme delta T lymphocytes, MAIT cells, Natural Killer T cells)

SECONDARY OUTCOMES:
UTC activation/inhibition profile | 18 months
  UTC activation/inhibition based on cell surface markers expression such as Cluster of Differenciation (CD) 69 and Programmed cell death 1 (PD-1)
UTC production of pro-inflammatory cytokines | 18 months
  Analysis of the level of IL-17, Interferon γ (IFNγ) and Tumor Necrosis Factor α (TNFα) produced by UTC
UTC capacity to mediate cytotoxicity | 18 months
  UTC cytotoxic profile based on Granzyme B and Cluster of Differenciation (CD) 107a expression

CONTACTS AND LOCATIONS:
Overall Officials: Youenn JOUAN, MD, Principal Investigator — University Hospital, Tours
Locations (2):
- France (2):
  - Cystic Fibrosis Resource and Competence Center, University Hospital, Tours, Tours
  - Pulmonology Department, University Hospital, Tours, Tours

IPD SHARING:
Plan to Share IPD: Undecided